CLINICAL TRIAL: NCT06862011
Title: Evaluation of Structured Sexual Health Counseling for Primiparous Pregnant Women Based on PLISSIT Model Supported by Motivational Interviewing
Brief Title: Evaluation of Sexual Health Counseling for Primiparous Pregnant Women Using PLISSIT Model and Motivational Interviewing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Özlem SEYMEN, Tokat Gaziosmanpasa University, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU-OS
Record Dates: First submitted 2025-02-10; First posted 2025-03-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; PLISSIT Model; Primiparity
Keywords: pregnancy; primiparous; PLISSIT; Sexual counseling
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant, Outcomes Assessor
Masking Description: The data from the study will be examined by an independent statistician. The person doing the analysis will not know the groups. Pregnant women included in the study will later learn which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (pregnant women receiving sexual counselling) (Experimental): In the intervention phase of the study, sexual counseling based on the PLISSIT model supported by motivational interviewing will be provided. The average duration of each counseling session is planned to be 60 minutes.
  Interventions: Behavioral: control group
- Control Group (pregnant women not receiving sexual counselling) (No Intervention): Scales and forms for the control group will be completed at the end of the second and fourth weeks.

INTERVENTIONS:
Behavioral: control group — Only surveys will be filled out.
  Arms: Intervention group (pregnant women receiving sexual counselling)

SUMMARY:
This study is a simple randomized controlled intervention study to evaluate the effects of sexual counseling given to primiparous pregnant women using motivational interviewing on sexual self-efficacy, attitude towards sexuality and quality of sexual life.

HO: There is no difference between the mean Sexual Function Scale score in the last evaluation of pregnant women in the intervention and control groups.

H0a: There is no difference between the mean Sexual Self-Efficacy Scale score in the last evaluation of pregnant women in the intervention and control groups.

H0b: There is no difference between the mean Attitude Towards Sexuality During Pregnancy Scale score in the last evaluation of pregnant women in the intervention and control groups.

H0c: There is no difference between the mean Sexual Life Quality Scale score in the last evaluation of pregnant women in the intervention and control groups.

DETAILED DESCRIPTION:
Pregnancy is a natural process that involves hormonal, physical, and social changes, affecting a woman's mood, relationships, and sexual life. The first pregnancy is a significant transition period, during which women may experience various fears related to sexuality, such as fear of miscarriage, premature birth, harming the baby, or increased risk of infection. These concerns often lead to a decrease in sexual activity during pregnancy.

The PLISSIT Model is suggested as an effective approach for assessing sexual health during pregnancy. This model consists of four stages: permission for expressing thoughts and concerns about sexuality, providing limited information, offering specific suggestions, and referring to intensive therapy when necessary. Additionally, the motivational interviewing method can help pregnant individuals recognize conflicting emotions and make positive behavioral changes.

Research indicates that sexual knowledge impacts sexual function, and participation in educational programs can improve sexual health during pregnancy. However, studies also show that healthcare professionals often lack sufficient support in this area. Nurses play a crucial role in educating and counseling pregnant women to enhance their awareness of sexual health. The absence of sexual health recommendations in the Ministry of Health's prenatal care guidelines highlights a gap in this area. Improving sexual quality of life during pregnancy is essential for strengthening women's self-confidence and sense of adequacy.

In the study, the data collection tools used were the **Inclusion Criteria Questionnaire (ICQ), Personal Information Form, Sexuality Diary, Female Sexual Function Index (FSFI), Sexual Self-Efficacy Scale (SSES), Attitudes Towards Sexuality During Pregnancy Scale (ATSPS), and Sexual Quality of Life Questionnaire-Female Version (SQOL-F).**

* **ICQ:** A ten-item form assessing the eligibility criteria for pregnant participants. Women who scored below 26.55 on the FSFI and answered all questions as "yes" were included in the study.
* **Personal Information Form:** A 15-item form assessing the socio-demographic and obstetric characteristics of pregnant individuals.
* **FSFI:** A scale evaluating female sexual function. A score below 26.55 indicates female sexual dysfunction.
* **SSES:** A scale measuring individuals' sexual self-efficacy, ranging from 0 to 40. Higher scores indicate higher sexual self-efficacy.
* **ATSPS:** A 34-item Likert-type scale assessing attitudes toward sexuality during pregnancy. Higher scores indicate a more positive attitude. The cutoff point is set at 111.5.

ELIGIBILITY:
Inclusion Criteria:

* Those over 19 years of age
* Those in their first pregnancy
* Those in their 8th-16th weeks of pregnancy
* Those who are sexually active
* Those who have a score of less than 26.55 on the Female Sexual Function Scale (FSFI)

Exclusion Criteria:

* Those who have given birth prematurely
* Those who have developed a pregnancy complication that prevents coitus at any stage of the study (placenta previa, preterm premature rupture of membranes)
* Those who do not comply with the study plan
* Those who have received any sexual counseling
* Those who have experienced a life crisis (death of partner, divorce, moving, etc.)
* Those who want to withdraw from the study at any stage of the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Scale | 5 weeks
  The Female Sexual Function Scale will be used to evaluate the sexual functions of pregnant women. The total score that can be obtained from the scale is between a minimum of 2 and a maximum of 36 points. Increasing scores indicate a good level of sexual function. If the total KCFI score is 30 and above, the sexual function level is defined as "good", between 23-29 points as "medium", and less than 23 points as low, and the cut-off value of the scale is 26.55. A total KCFI score of 26.55 and below indicates that the level of sexual function is inadequate.

SECONDARY OUTCOMES:
Sexual Self-Efficacy Scale | 5 weeks
  will be used to determine the sexual self-efficacy levels of pregnant women. The scale is one-dimensional. The lowest score that can be obtained from the scale is 0, the highest score is 40. High scores indicate a high level of sexual self-sufficiency belief.

OTHER OUTCOMES:
Attitude Towards Sexuality During Pregnancy Scale ( | 5 weeks
  It will be used to evaluate pregnant women's attitudes towards sexuality during pregnancy. The lowest possible total score from the Attitudes Towards Sexuality During Pregnancy Scale was calculated as 34 and the highest as 170. An increase in the total score from the GCCTS indicates that attitudes towards sexuality during pregnancy are positive, while a decrease in the total score indicates that attitudes towards sexuality during pregnancy are negative.
Sexual Life Quality Scale-Female Version | 5 weeks
  It will be used to evaluate the Sexual Life Quality of pregnant women. The range of scores that can be obtained from this scale varies between 18-100. Before calculating the total score of the scale, the scores of items 1, 5, 9, 13, 18 must be reversed. Increasing scores from the scale indicate that the quality of sexual life has also increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting information: CSR
Supporting Information: CSR